CLINICAL TRIAL: NCT00005366
Title: Biobehavioral Mechanisms of Blood Pressure Regulation
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4253; R01HL049427 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2001-04

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension

SUMMARY:
To investigate the role of biobehavioral factors in the pathogenesis of concentric left ventricular hypertrophy.

DETAILED DESCRIPTION:
BACKGROUND:

Hypertension is more prevalent in Black than white men, and is more prevalent in men than women. Furthermore, even controlling for blood pressure, concentric left ventricular hypertrophy, an early structural adaptation of hypertension, is more prevalent in Black than white men, and more prevalent in men than women. Concentric left ventricular hypertrophy is the strongest predictor, other than age, of the cardiovascular morbidity associated with high blood pressure.

DESIGN NARRATIVE:

In a biracial sample, concentric left ventricular hypertrophy and concentric remodelling were assessed by echocardiographic measures of left ventricular mass and relative wall thickness. Laboratory procedures were used to: (i) assess hemodynamic and neurohumoral responses during exposure to a diverse battery of physical and psychological stressors, and; (ii) evaluate alpha and beta adrenergic receptor responsiveness, baroreceptor reflex gain and minimal forearm vascular resistance. Since blood pressure during a typical workday was an established predictor of left ventricular hypertrophy, it was also assessed. A new biobehavioral model was tested that implicated the hemodynamic pattern of behaviorally-evoked pressor responses in the pathogenesis of concentric left ventricular hypertrophy. One prediction of this model was that a predisposition to exhibit increased vascular resistance during stress (characteristic of black men) would favor the development of concentric hypertrophy. Thus, systemic vascular resistance responses, evaluated in the laboratory, were hypothesized to independently predict left ventricular mass and relative wall thickness, even after controlling for established risk factors, including workday blood pressure. Sympathetic nervous system function was examined to test hypothesized mechanisms responsible for race and gender differences in the hemodynamic patterns of blood pressure regulation. The results of these studies emphasized the importance of race and gender in prescribing pharmacological and/or behavioral treatment for hypertensive heart disease.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Ages: 25 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 1993-09; Study Completion 1998-08 (Actual)

REFERENCES:
- [Background] Watkins LL, Grossman P, Sherwood A. Noninvasive assessment of baroreflex control in borderline hypertension. Comparison with the phenylephrine method. Hypertension. 1996 Aug;28(2):238-43. doi: 10.1161/01.hyp.28.2.238. PMID 8707388
- [Background] Sherwood A, May CW, Siegel WC, Blumenthal JA. Ethnic differences in hemodynamic responses to stress in hypertensive men and women. Am J Hypertens. 1995 Jun;8(6):552-7. doi: 10.1016/0895-7061(95)00036-O. PMID 7662238
- [Background] Blumenthal JA, Thyrum ET, Gullette ED, Sherwood A, Waugh R. Do exercise and weight loss reduce blood pressure in patients with mild hypertension? N C Med J. 1995 Feb;56(2):92-5. PMID 7898595
- [Background] Sherwood A, Hinderliter AL, Light KC. Physiological determinants of hyperreactivity to stress in borderline hypertension. Hypertension. 1995 Mar;25(3):384-90. doi: 10.1161/01.hyp.25.3.384. PMID 7875764
- [Background] Carels RA, Blumenthal JA, Sherwood A. Emotional responsivity during daily life: relationship to psychosocial functioning and ambulatory blood pressure. Int J Psychophysiol. 2000 Apr;36(1):25-33. doi: 10.1016/s0167-8760(99)00101-4. PMID 10700620
- [Background] Sherwood A, Johnson K, Blumenthal JA, Hinderliter AL. Endothelial function and hemodynamic responses during mental stress. Psychosom Med. 1999 May-Jun;61(3):365-70. doi: 10.1097/00006842-199905000-00017. PMID 10367618
- [Background] Carels RA, Szczepanski R, Blumenthal JA, Sherwood A. Blood pressure reactivity and marital distress in employed women. Psychosom Med. 1998 Sep-Oct;60(5):639-43. doi: 10.1097/00006842-199809000-00022. PMID 9773771
- [Background] Watkins LL, Grossman P, Krishnan R, Sherwood A. Anxiety and vagal control of heart rate. Psychosom Med. 1998 Jul-Aug;60(4):498-502. doi: 10.1097/00006842-199807000-00018. PMID 9710297
- [Background] Carels RA, Sherwood A, Blumenthal JA. Psychosocial influences on blood pressure during daily life. Int J Psychophysiol. 1998 Mar;28(2):117-29. doi: 10.1016/s0167-8760(97)00090-1. PMID 9545650
- [Background] Carels RA, Sherwood A, Szczepanski R, Blumenthal JA. Ambulatory blood pressure and marital distress in employed women. Behav Med. 2000 Summer;26(2):80-5. doi: 10.1080/08964280009595755. PMID 11147293